CLINICAL TRIAL: NCT03060590
Title: Association of Uremic Toxins and Sacropenia in Hemodialysis Patients
Brief Title: Roles of Uremic Toxins in Uremic Sacropenia
Status: Completed | Type: Observational
Sponsor: Tungs' Taichung Metroharbour Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 105055
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Sarcopenia
Keywords: sarcopenia, uremic toxins
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background. In advanced chronic kidney disease (CKD), multiple metabolic and nutritional abnormalities may contribute to the impairment of skeletal muscle mass and function thus predisposing patients to the condition of sarcopenia. Herein, we aim to investigate the association of uremic toxins and sacropenia. In addition, the prevalence and mortality predictive power of sarcopenia, defined by different methods, in a cohort of hemodialysis patients.

Methods. We plan to evaluate 300 HD patients. Sarcopenia was defined as reduced muscle function assessed by handgrip strength (HGS <30th percentile of a population-based reference adjusted for sex and age) plus diminished muscle mass assessed by different methods: (i) midarm muscle circumference (MAMC) <90% of reference value (A), (ii) muscle wasting by DEXA (B) and (iii) reduced skeletal muscle mass index (<10.76 kg/m² men; <6.76 kg/m² women) estimated by bioelectrical impedance analysis (BIA) (C). Serum levels of 3 established uremic toxins such as indoxyl sulfate, p-cresol and hippuric acid will be measured. Besides, various relevant inflammatory markers will also be assessed. Patients will be followed for up to 3 years for all-cause mortality.

DETAILED DESCRIPTION:
Patients and Methods

This study will included 300 consecutive patients receiving maintenance hemodialysis at the outpatient dialysis center of the Tungs Taichung Metroharbour Hospital, Taichung Taiwan. Recruitment will start after approval of the Ethics Committee of our hospital. Exclusion criteria were age of <20 and >90 years, clinical signs of acute infection during the month preceding the inclusion, active cancer or liver disease at the time of evaluation, previous diagnosis of immunological diseases and unwillingness to participate in the study. Physician will perform a complete chart review and interviewed each patient regarding their clinical history.

All MHD patients enrolled in our study will be tested with DEXA and bioelectrical impedance analysis (BIA) and grip strength. Demographic data was collected and anthropometric measurement such as mid-arm muscle circumference (MAMC) calf circumference, and laboratory examination are conducted.

Handgrip strength

Muscle strength is assessed in the dominant hand using a Jamar hand dynamometer (Lafayette Instrument Company, USA). Patients are ﬁrst familiarized with the device and were then examined standing with both arms extended sideways from the body with the dynamometer facing away from the body. Patients were instructed to grip the dynamometer with the maximum strength in response to a voice command, and the highest value of three measurements was considered for the study. Handgrip strength (HGS) values under the 30th percentile from a speciﬁc-population reference value adjusted for age and sex were considered as reduced.

Anthropometry

Body mass index (BMI) is calculated as weight in kilograms divided by height in squared meters. MAMC is calculated according to the following equation, based on mid-arm circumference (measured at mid-point from the acromion to olecranon) and the triceps skinfold (using caliper Lange®, Cambridge Scientiﬁc Industries, Inc.).

Values of MAMC were compared with the 50th percentile of NHANES II and standard adequacy of <90% was considered as reduced muscle mass .

Bioelectrical impedance analysis

Body composition was measured using an 8-contact electrode bioelectrical impedance analysis (BIA) device (Tanita BC-418, Tanita, Tokyo, Japan), and followed the standard procedure and the manufacturer's instructions. This BIA device was used to measure the whole body and segmental impedance (± 1Ω) at a frequency of 50 kHz, and it provided valid muscle mass estimates (kg) of each of the four extremities.[2 Appendicular muscle mass (ASM) was calculated as the sum of the estimated muscle mass for the arms and legs. A relative skeletal muscle mass index (ASM/ht2) normalized for height was defined as the ratio of ASM (kg) and the height squared(m2). For this analysis, we defined muscle mass cut-off points according to the distribution of ASM/ht2 of a young population comprising 998 healthy adults (aged 20-40 years) or the study population. A participant was considered to have low muscle mass if his or her ASM/ht2 was below -2 standard deviations of the reference young adult values defined in previous studies (6.76 kg/m2 for men and 5.28 kg/m2 for women).

Sarcopenia diagnosis

The diagnosis of sarcopenia was based on the presence of derangements in both muscle function and muscle mass. For the purpose of the study, we considered one muscle function indicator (reduced HGS) associated with one of three indicators of muscle mass (MAMC, DEXA or BIA). Therefore, reduced HGS in association with an MAMC of <90% of the standard adequacy (Method A), presence of muscle wasting by DEXA (MethodB) or reduced SMMI by BIA(MethodC) were considered as diagnosis of sarcopenia.

Laboratorial parameters

All blood samples are collected during the midweek dialysis from the AV fistula, immediately after the insertion of the dialysis cannula but before the administration of heparin. Blood is sampled in 4 c.c. Venoject II tubes, centrifuged (10 min, 3000 rpm) and immediately store at -70°C until assayed. Serum albumin, urea, creatinine, and total protein concentrations in serum are determined according to standard methods. The serum levels of hsCRP are measured using a Behring Nephelometer II (Dade Behring, Tokyo, Japan). Serum concentrations of total p-cresol sulfate, hippuric acid and IS (i.e., combined free and protein bound fractions) are analyzed with High-performance liquid chromatography (HPLC). Briefly, for binding competition, 200μl serum to which we added 20μl 0.50mM 1-naphthalenesulfonic acid (internal standard) was vortex-mixed with 250μl 0.24M sodium octanoate (binding competitor).After incubation at room temperature for 5min, we added 2ml cold acetone to precipitate proteins. Following vortex-mixing and centrifuging at 4 ◦C, 1860×g for 20 min, the supernatant was transferred to 12mm×100mm, GL 14 glass test tubes and 2ml dichloromethane was added. After vortex-mixing and centrifuging at 4 ◦C, 1860×g for 10min, 200μl of the upper layer was transferred to glass autosampler vials, followed by addition of 20μl 1M HCl and 15μl was injected onto the HPLC. The HPLC analysis was performed on an Agilent 1100 series LC (Santa Clara, CA),and Agilent ChemStations software were used for the chromatographic analysis. The separation was carried out on a ZORBAX SB-C18 Solv Saver Plus HPLC column (5 μm, 3.0 mm×150 mm).at a flow rate of 0.6 ml/min. Mobile phase A is 0.2% trifluoroacetic acid in Milli-Q water and mobile phase B is 0.2% trifluoroacetic acid in acetonitrile. The analytical method consists of an isocratic run with 92% mobile phase A for 23 min.. Each analytical run was followed by a 1.3 min washout gradient to 100% B. Column temperature was 25 ◦C, and autosampler tray temperature was 6 ◦C. We quantified the analytes by using the analyte to standard peak area ratio on a Agilent 1100 High Performance Fluorescence detector G1321A and Agilent 1100 Series UV-Visible detectors G1314A. Detector settings were λex 260 nm/λem288nm for p-cresyl sulfate and λex 280 nm/λem 390nm for indoxyl sulfate and internal standard. Hippuric acid was monitored by UV-Vis detector at 254 nm. Quantitative results are obtained and calculated in terms of their concentrations (mg/L).

Blood samples are also collected before dialysis for measurement of oxidative stress (CML, Nε-(carboxymethyl)lysine ) and inflammatory markers (IL-6). Serum Nε-(carboxymethyl)lysine (CML) was determined using enzyme-linked immunosorbent assay (R&D system, Minneapolis, MN, USA). Similarly, the concentration of IL-6 is also assessed using Quantikine Human Interleukin Immunoassay (R&D Systems Minneapolis, MN, USA) with a detection limit of 15 pg/L and 0.12 pg/mL, respectively. In addition, serum irisin, urotensin II, follistatin and alpha 1 antichymotrypsin concentrations are measured by using the human enzyme-linked immunosorbent assay (ELISA) kits in accordance with the manufacturer's instructions. The All determinations are performed in duplicate, and the mean value is used.

Statistical analyses

The variables are expressed in mean±SD, median (interquartile range) or proportions. Variable distributions are tested by e.g. Shapiro Wilk test, and those not normally distributed are standardized by using z-score.Studentt-test or Chi-square test is employed for the comparisons between sarcopenic and non-sarcopenic patients. Kappa test is used to evaluate the agreement among the methods. Survival analyses are made with the Kaplan-Meier survival curve and the Cox proportional hazard model. The univariate and multivariate Cox-regression analyses are presented as hazard ratio [HR; 95% conﬁdence intervals (CI)]. Statistical signiﬁcance is set at the level of P<0.05, and the analyses are performed by using the SPSS software version 18 (SPSS, Inc., Chicago, IL, USA)

ELIGIBILITY:
Inclusion Criteria:

* Both sexes aged between 20-90 years. Received stable hemodialysis at least 3 months. Written informed consent.

Exclusion Criteria:

* clinical signs of acute infection during the month preceding the inclusion, active cancer or liver disease at the time of evaluation, previous diagnosis of immunological diseases and unwillingness to participate in the study.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hemodialysis (HD) patients
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Presence of Sarcopenia | 3 years
  To evaluate the association of sacropenia defined according to 1. Low muscle mass 2. Low muscle strength 3. Low physical performance and serum levels of some uremic toxins such as indoxyl sulfate, p-cresol and hippuric acid will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Paik Seong Lim, PhD, Principal Investigator — Tungs' Taichung Metroharbour Hospital
Locations (1):
- Tungs' Taichung MetroHarbour Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No